CLINICAL TRIAL: NCT07021482
Title: Ultrasonographic Assessment of Airway Edema Induced by Intra-abdominal Pressure During Laparoscopic Cholecystectomy: A Prospective, Double-Blind, Randomized Study
Brief Title: Ultrasound Assessment of Airway Edema During Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Engin Çetin (Other Government)
Responsible Party: Sponsor-Investigator, Engin Çetin, Principal Investigator, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KSH-ANREA-EC-01
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Airway Edema; Perioperative Complication; Pneumoperitoneum
Keywords: Airway Ultrasound; Upper Airway Edema; Pneumoperitoneum; Intra-abdominal Pressure
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mmHg Pneumoperitoneum (Active Comparator): Patients in this group will undergo laparoscopic cholecystectomy with pneumoperitoneum maintained at 10 mmHg.
  Interventions: Diagnostic Test: 10 mmHg Pneumoperitoneum
- 14 mmHg Pneumoperitoneum (Active Comparator): Patients in this group will undergo laparoscopic cholecystectomy with pneumoperitoneum maintained at 14 mmHg.
  Interventions: Diagnostic Test: 14 mmHg Pneumoperitoneum

INTERVENTIONS:
Diagnostic Test: 10 mmHg Pneumoperitoneum — Laparoscopic cholecystectomy will be performed with intra-abdominal pressure maintained at 10 mmHg during insufflation. Standard anesthesia and surgical protocols will be followed.
  Arms: 10 mmHg Pneumoperitoneum
Diagnostic Test: 14 mmHg Pneumoperitoneum — Laparoscopic cholecystectomy will be performed with intra-abdominal pressure maintained at 14 mmHg during insufflation. Standard anesthesia and surgical protocols will be followed.
  Arms: 14 mmHg Pneumoperitoneum

SUMMARY:
This prospective, double-blind, randomized clinical trial aims to investigate the development of airway edema associated with intra-abdominal pressure during laparoscopic cholecystectomy. A total of 66 adult patients undergoing elective laparoscopic cholecystectomy under general anesthesia will be randomly assigned into two equal groups (33 patients per group) based on intra-abdominal pressure levels: low-pressure and standard-pressure pneumoperitoneum. Ultrasonographic measurements will be used to assess airway soft tissue thickness at predefined time points before and after the pneumoperitoneum. The primary objective is to determine whether increased intra-abdominal pressure contributes to postoperative airway edema, which may pose a risk during extubation.

DETAILED DESCRIPTION:
Airway edema can lead to difficult extubation and perioperative complications. Pneumoperitoneum during laparoscopic surgery increases intra-abdominal pressure (IAP), which may contribute to airway soft tissue edema due to cephalad fluid shifts and venous congestion. This prospective, randomized, double-blind study aims to assess whether different levels of IAP have a measurable effect on airway soft tissue thickness.

Patients aged 18 to 65 years, classified as ASA I-II, and scheduled for elective laparoscopic cholecystectomy will be included in the study. Upon arrival in the operating room, standard monitoring will be applied, anesthesia will be induced using intravenous sedation, and endotracheal intubation will be performed.

In the preoperative period, airway ultrasonography will be used to measure tongue thickness, midsagittal tongue cross-sectional area, tongue width, lateral pharyngeal wall thickness, parapharyngeal area thickness, and submental area thickness.

Patients will be randomly assigned into two groups:

Group 1: Patients receiving 10 mmHg intra-abdominal pressure Group 2: Patients receiving 14 mmHg intra-abdominal pressure

T0: Before intubation

T1: After intubation

T2: 30 minutes after the initiation of pneumoperitoneum

T3: 5 minutes after extubation

T4: 1 hour after extubation

T5: 2 hours after extubation

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* ASA physical status I-II
* Body mass index (BMI) < 30 kg/m²
* Mallampati score I-II
* Scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

* History of difficult intubation
* Upper respiratory tract infection
* Obstructive sleep apnea or STOP-Bang score ≥3
* Severe cardiopulmonary disease
* Pregnancy
* Indication for emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2025-06-18 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Lateral Pharyngeal Wall Thickness Measured by Airway Ultrasound | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (10 mmHg vs. 14 mmHg) on upper airway edema during laparoscopic cholecystectomy. The degree of airway edema will be assessed by measuring changes in lateral pharyngeal wall thickness using ultrasound before and after the procedure.

SECONDARY OUTCOMES:
ultrasonographic airway parameter -tongue width | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (10 mmHg vs. 14 mmHg) on upper airway edema during laparoscopic cholecystectomy. The degree of edema will be evaluated by changes in ultrasonographic measurements of upper airway structures (e.g., tongue thickness, midsagittal cross-sectional area, pharyngeal wall thickness) before and after the procedure.
ultrasonographic airway parameter -tongue volume | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (10 mmHg vs. 14 mmHg) on upper airway edema during laparoscopic cholecystectomy. The degree of edema will be evaluated by changes in ultrasonographic measurements of upper airway structures (e.g., tongue thickness, midsagittal cross-sectional area, pharyngeal wall thickness) before and after the procedure.
ultrasonographic airway parameter-pharyngeal thickness | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (10 mmHg vs. 14 mmHg) on upper airway edema during laparoscopic cholecystectomy. The degree of edema will be evaluated by changes in ultrasonographic measurements of upper airway structures (e.g., tongue thickness, midsagittal cross-sectional area, pharyngeal wall thickness) before and after the procedure.
ultrasonographic airway parameter- neck circumference | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To compare the effect of two different pneumoperitoneum pressures (10 mmHg vs. 14 mmHg) on upper airway edema during laparoscopic cholecystectomy. The degree of edema will be evaluated by changes in ultrasonographic measurements of upper airway structures (e.g., tongue thickness, midsagittal cross-sectional area, pharyngeal wall thickness) before and after the procedure.
oxygen saturation changes | Immediately after extubation and during early recovery (within the first 2 hours postoperative)
  To evaluate the clinical impact of pneumoperitoneum pressure (10 mmHg vs. 14 mmHg) on postoperative airway outcomes. Clinical indicators such as oxygen saturation changes, signs of airway obstruction, hoarseness, sore throat, hypoxia, stridor, and re-intubation will be recorded. The incidence of these complications will be compared between groups to assess whether higher pressure is associated with increased airway-related morbidity.
hoarseness | Immediately after extubation and during early recovery (within the first 2 hours postoperative)
  To evaluate the clinical impact of pneumoperitoneum pressure (10 mmHg vs. 14 mmHg) on postoperative airway outcomes. Clinical indicators such as oxygen saturation changes, signs of airway obstruction, hoarseness, sore throat, hypoxia, stridor, and re-intubation will be recorded. The incidence of these complications will be compared between groups to assess whether higher pressure is associated with increased airway-related morbidity.
stridor | Immediately after extubation and during early recovery (within the first 2 hours postoperative)
  To evaluate the clinical impact of pneumoperitoneum pressure (10 mmHg vs. 14 mmHg) on postoperative airway outcomes. Clinical indicators such as oxygen saturation changes, signs of airway obstruction, hoarseness, sore throat, hypoxia, stridor, and re-intubation will be recorded. The incidence of these complications will be compared between groups to assess whether higher pressure is associated with increased airway-related morbidity.
re-intubation | Immediately after extubation and during early recovery (within the first 2 hours postoperative)
  To evaluate the clinical impact of pneumoperitoneum pressure (10 mmHg vs. 14 mmHg) on postoperative airway outcomes. Clinical indicators such as oxygen saturation changes, signs of airway obstruction, hoarseness, sore throat, hypoxia, stridor, and re-intubation will be recorded. The incidence of these complications will be compared between groups to assess whether higher pressure is associated with increased airway-related morbidity.
sore throat | Immediately after extubation and during early recovery (within the first 2 hours postoperative)
  To evaluate the clinical impact of pneumoperitoneum pressure (10 mmHg vs. 14 mmHg) on postoperative airway outcomes. Clinical indicators such as oxygen saturation changes, signs of airway obstruction, hoarseness, sore throat, hypoxia, stridor, and re-intubation will be recorded. The incidence of these complications will be compared between groups to assess whether higher pressure is associated with increased airway-related morbidity.
Correlation Between Intravenous Fluid Volume and Airway Edema | T0: Before intubation T1: After intubation T2: 30 minutes after the initiation of pneumoperitoneum T3: 5 minutes after extubation T4: 1 hour after extubation T5: 2 hours after extubation
  To evaluate the correlation between the total intravenous fluid volume administered intraoperatively and the degree of airway edema, as measured by changes in ultrasonographic airway parameters (e.g., tongue thickness, pharyngeal wall thickness) at defined time points.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aytac BG, Soyal OB. Ultrasonographic evaluation of the postoperative airway edema after robotic prostatectomy: a single center observational study. Eur Rev Med Pharmacol Sci. 2023 Sep;27(18):8505-8513. doi: 10.26355/eurrev_202309_33775. PMID 37782166